CLINICAL TRIAL: NCT00908947
Title: CONTINuous Infra-Inguinal Stenting Using the Bard® LifeStent® VascUlar Stent SysteMs ("CONTINUUM")
Acronym: CONTINUUM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll the required number of subjects
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-08-001
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Results first posted 2019-11-06 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Superficial Femoral Artery Stenosis
Keywords: SFA; Stent; Popliteal; infrainguinal; LifeStent; Peripheral; Arterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Overall Study (Experimental): PTA plus stenting with the LifeStent® Vascular Stent System
  Interventions: Device: PTA followed by placement of LifeStent® Vascular Stent

INTERVENTIONS:
Device: PTA followed by placement of LifeStent® Vascular Stent — PTA followed by placement of LifeStent® Vascular Stent
  Other Names: LifeStent® Vascular Stent; LifeStent® XL Vascular Stent; LifeStent® SOLO(TM) Vascular Stent

SUMMARY:
The objectives of this study are to collect post-market confirmatory evidence of the safety and effectiveness of the Bard® LifeStent® Vascular Stent System and LifeStent® XL Vascular Stent System (together the "LifeStent® Vascular Stent System").

DETAILED DESCRIPTION:
The study is a prospective, multi-center, single-arm, non-randomized study enrolling up to 234 subjects with lifestyle-limiting claudication or ischemic rest pain attributable to lesion(s) (stenosed, occluded, restenosed, or re-occluded) in the infra-inguinal segment (Superficial femoral artery [SFA] and/or proximal popliteal artery) that are amenable to treatment by percutaneous transluminal angioplasty (PTA) and stenting. All subjects enrolled in the study will receive PTA and stenting.

ELIGIBILITY:
Inclusion Criteria:

1. The subject provides written informed consent using an Informed Consent Form (ICF) that is reviewed and approved by the Institutional Review Board (IRB) for the site.
2. Subject agrees to comply with the protocol-mandated follow-up procedures and visits.
3. The subject is ≥ 21 years old.
4. Male or female subjects; female subjects of childbearing potential must have a negative urine pregnancy test at the time of screening.
5. The subject has lifestyle-limiting claudication or ischemic rest pain defined as: Rutherford Category 2-4.
6. The target lesion(s) has angiographic evidence of stenosis or restenosis ≥ 50% or occlusion (by visual estimate) and is amenable to PTA with stenting.
7. The total target lesion(s) length must be ≤ 240 mm.
8. The target vessel reference diameter is ≥ 4.0 mm and ≤ 6.5 mm (by visual estimate), and therefore appropriate for treatment with available stent diameters of 6.0 mm and 7.0 mm.

Exclusion Criteria:

1. The subject is unable or unwilling to provide informed consent, or is unable or unwilling to conform to the study protocol follow-up procedures and visits.
2. The subject has claudication or critical limb ischemia described as Rutherford Category 1 (mild claudication), 5 (minor tissue loss) or 6 (major tissue loss.
3. The subject has multiple stenoses or occlusions > 240 mm.
4. The subject has a previous stent or stent graft located in the target vessel.
5. The subject has flow-limiting stenosis or occlusion of the inflow tract that cannot be adequately corrected (≤ 30% residual stenosis) prior to treatment of the target lesion(s). Investigator standard of care practices shall be utilized for treatment of inflow.
6. The subject has a known contraindication (including allergic reaction) to antiplatelet/anticoagulant medications, nickel, titanium, tantalum or sensitivity.
7. The subject has a known contraindication to contrast media that is not amenable to pretreatment with steroids or/and antihistamines.
8. The subject has a known history of bleeding diatheses or coagulopathy.
9. The subject has concomitant renal failure with a creatinine of > 2.5 mg/dL.
10. The subject is currently on dialysis or receiving systemic immunosuppressive therapy.
11. The subject has known concomitant hepatic insufficiency, thrombophlebitis, uremia, systemic lupus erythematosus, septicemia or deep vein thrombosis at the time of the index procedure.
12. The subject is currently participating in an investigational drug or another investigational device study that has not completed the primary endpoint, or that clinically interferes with the study endpoints. Note: trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
13. The subject has another medical condition, which, in the opinion of the Investigator, may cause him/her to be non-compliant with the protocol, confound the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of study procedures and follow-up.
14. The subject has extensive peripheral vascular disease, which in the opinion of the Investigator, would preclude safe insertion of an introducer sheath.
15. The target lesion(s) is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion(s).
16. There is angiographic evidence of unresolved thrombus at the target lesion(s) or within the target vessel that does not resolve with infusion of thrombolytics and/or mechanical thrombectomy (using an approved device) without adverse events/complications.
17. The subject has undergone any non-iliac percutaneous intervention(s) < 7 days prior to the index procedure.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2011-02; Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey P Carpenter, MD, Principal Investigator — The Cooper Health System; Mark D Mewissen, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (29):
- United States (29):
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Mission Cardiovascular Research Institute, Pleasanton, California
  - South Florida Medical Imaging, PA, Fort Lauderdale, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Loyola University Chicago, Chicago, Illinois
  - Heartland Vascular Center, Joliet, Illinois
  - Prairie Education and Research Cooperative (PERC), Springfield, Illinois
  - Cardiovascular Research of Northwest Indiana, LLC., Munster, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Kentucky Heart Foundation, Ashland, Kentucky
  - Steward St. Elizabeth Medical Center of Boston Inc., Boston, Massachusetts
  - Metropolitan Hospital d/b/a Metro Health Hospital, Wyoming, Michigan
  - Midwest Aortic Vascular Institute P.C, North Kansas City, Missouri
  - The Cooper Health System, Camden, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - The Huntington Heart Center, Huntington, New York
  - Saint Vincent Consultants in Cardiovascular Diseases, LLC, Erie, Pennsylvania
  - Trustees of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - PinnacleHealth Cardiovascular Institute, Wormleysburg, Pennsylvania
  - South Carolina Heart Center, P.A., Columbia, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Sanford Research, Sioux Falls, South Dakota
  - University Surgical Associates, LLC, Chattanooga, Tennessee
  - BCS Heart, LLP., College Station, Texas
  - Houston Center for Vascular Health, Houston, Texas
  - The Methodist Hospital Research Institute dba Houston Methodist Research Institute, Houston, Texas
  - Aurora Medical Group, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled on February 9, 2011 and the final follow-up was completed on September 19, 2018.
Groups:
- LifeStent: Percutaneous Transluminal Angioplasty (PTA) followed by placement of LifeStent® Vascular Stent: PTA followed by placement of LifeStent® Vascular Stent
Period: Overall Study
Arm/Group | LifeStent
Started | 173
Completed | 83
Not Completed | 90

BASELINE CHARACTERISTICS:
Groups:
- LifeStent: Percutaneous trasluminal angioplasty (PTA) plus stenting with the LifeStent® Vascular Stent System
  PTA followed by placement of LifeStent® Vascular Stent: PTA followed by placement of LifeStent® Vascular Stent
Arm/Group | LifeStent
Number analyzed (Participants) | 173
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 158
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 22
  White | 138
  More than one race | 1
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 173
Rutherford Category [Count of Participants; unit: Participants] — Population: data was collected for 171 out of 173 patients, thus, 2 patients did not have Rutherford category assigned at baseline.
  Participants
    0: Asymptomatic: number analyzed (Participants) | 171
    0: Asymptomatic | 0
    1: Mild Claudication: number analyzed (Participants) | 171
    1: Mild Claudication | 0
    2: Moderate Claudication: number analyzed (Participants) | 171
    2: Moderate Claudication | 25
    3: Severe Claudication: number analyzed (Participants) | 171
    3: Severe Claudication | 114
    4: Ischemic Rest Pain: number analyzed (Participants) | 171
    4: Ischemic Rest Pain | 31
    5: Minor Tissue Loss: number analyzed (Participants) | 171
    5: Minor Tissue Loss | 0
    6: Major Tissue Loss: number analyzed (Participants) | 171
    6: Major Tissue Loss | 1
Number of Target Lesions per Subject [Count of Participants; unit: Participants]
  1 | 161
  2 | 10
  3 | 2
Target Limb [Count of Participants; unit: Participants]
  Left | 91
  Right | 82
Lesion Type [Number; unit: Lesion type]
  Stenosed | 124
  Occlusion | 57
  Restenosed | 6
Lesion Location [Number; unit: Lesions] — "Unknown category" includes 6 lesions for which anigiographic location data was not available pre-procedure.
  Lesions
    Proximal 1/3 of Superficial femoral Artery (SFA) | 32
    Distal 1/3 of Superficial femoral artery (SFA) | 80
    Mid 1/3 of Superficial femoral artery (SFA) | 69
    Unknown | 6
Lesion Calcification [Number; unit: Lesions]
  Absent | 25
  Mild | 54
  Moderate | 68
  Severe | 40
  Lesion Ulceration | 24
  Lesion Thrombus | 5

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: Freedom From Death at 30-days and 12-months Post-Index Procedure.
Description: Primary safety endpoint defined as freedom from occurrence of death at 30-days and 12-months post-index procedure.
Time Frame: 30-days and 12-months
Population: One subject expired on day 22 post-index procedure due to pneumonia (total N = 173, as per Participant Flow). The event was unrelated to study device but possibly related to procedure as adjudicated by the Clinical Events Committee (CEC).
Measure: Number (95% Confidence Interval); unit: Probability of Event Free
Arm/Group | Overall Study
Number analyzed (Participants) | 172
Probability of Event Free
  30-days Post Index Procedure | 0.994 [0.959 to 0.999]
  12-Months Post Index Procedure: number analyzed (Participants) | 149
  12-Months Post Index Procedure | 0.951 [0.904 to 0.975]

2. Primary Outcome: Primary Effectiveness Endpoint: Primary Target Lesion Patency (TLP) at Time of Procedure and 12-Months Post-Index Procedure
Description: The primary effectiveness endpoint of the study, device success, collectively measured both acute and chronic effectiveness.
  Acute effectiveness is defined as successful delivery of the stent to the intended site with the post-deployment stent length being within 10% of the pre-deployment stent length.
  Chronic effectiveness is defined as Primary Target Lesion Patency (TLP) at 12-months post-index procedure, as measured by Duplex Ultrasound (DUS).
Time Frame: At time of procedure (acute) and 12-months post-index procedure (Chronic)
Measure: Number (95% Confidence Interval); unit: Probability of effectiveness
Arm/Group | Overall Study
Number analyzed (Participants) | 173
Probability of effectiveness
  Acute effectiveness | 0.990 [0.948 to 1.000]
  Device success at 12-month | 0.727 [0.618 to 0.810]

3. Secondary Outcome: Freedom From Target Lesion Revascularization (TLR) and/or Target Vessel Revascularization (TVR) at 12-months Post-index Procedure.
Description: Target Lesion Revascularization (TLR) is defined as the interval following the index procedure until the first revascularization procedure of the target lesion. Target Vessel Revascularization (TVR) is defined as the interval following the index procedure until the first revascularization procedure (e.g. PTA, stenting, surgical bypass, etc.) in the target vessel.
Time Frame: 12-months post-index procedure
Measure: Number (95% Confidence Interval); unit: Probability of Event Free
Arm/Group | Overall Study
Number analyzed (Participants) | 173
Probability of Event Free | 0.822 [0.752 to 0.873]

4. Secondary Outcome: Primary Safety: Freedom From Death at 30-days and 12-months Post-Index Procedure for Target Lesion Lengths >160 mm Compared With LifeStent 200 mm.
Description: • Primary Safety (freedom from occurrence of death at 30-days and 12-months post-index procedure) of the Target Lesion Lengths > 160 mm subgroup compared to the Target Lesions treated with the 200 mm LifeStent® subgroup.
Time Frame: 30-days and 12-months Post -Index Procedure
Population: Target lesions >160mm = 18 participants, and Target lesions treated with 200mm LifeStent = 41 participants. Therefore N=59.
Measure: Number (90% Confidence Interval); unit: Probability of Event Free
Arm/Group | Overall Study
Number analyzed (Participants) | 59
Probability of Event Free
  Target Lesion Length > 160 at 30-days: number analyzed (Participants) | 17
  Target Lesion Length > 160 at 30-days | 1 [1.000 to 1.000]
  Target Lesion Length > 160 at 12-months: number analyzed (Participants) | 12
  Target Lesion Length > 160 at 12-months | 0.871 [0.641 to 0.958]
  Target Lesion Length 200 mm at 30-days: number analyzed (Participants) | 41
  Target Lesion Length 200 mm at 30-days | 1.000 [1.000 to 1.000]
  Target Lesion Length 200 mm at 12-months: number analyzed (Participants) | 39
  Target Lesion Length 200 mm at 12-months | 0.976 [0.880 to 0.995]

5. Secondary Outcome: Primary Effectiveness: Device Success at 12-Months Post-Index Procedure for Target Lesion Lengths > 160 mm Compared to LifeStent 200 mm.
Description: Primary Effectiveness (Device Success) of Target Lesion Lengths > 160 mm subgroup compared to the Target Lesions treated with the 200 mm LifeStent® subgroup.
Time Frame: 12-months Post-Index Procedure
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Probability Device Success
Groups:
- LifeStent: PTA plus stenting with the LifeStent® Vascular Stent System
  PTA followed by placement of LifeStent® Vascular Stent: PTA followed by placement of LifeStent® Vascular Stent
Arm/Group | LifeStent
Number analyzed (Participants) | 59
Probability Device Success
  Target Lesion Length > 160 at 12 months: number analyzed (Participants) | 18
  Target Lesion Length > 160 at 12 months | 0.438 [0.143 to 0.704]
  Target Lesion Length LifeStent 200 mm at 12 months: number analyzed (Participants) | 41
  Target Lesion Length LifeStent 200 mm at 12 months | 0.600 [0.399 to 0.753]

6. Secondary Outcome: Freedom From Fracture at 12 and 24-Months Post-Index Procedure
Description: Freedom from Fracture (FFF) at 12- and 24-months post-index procedure.
Time Frame: 12- and 24-months post-index procedure
Population: The results presented in this analysis include active patients that had available x-ray images appropriate for analysis by the core-lab at follow-up time (12 and 24 months). Therefore n=166 instead of N=173.
Measure: Number (90% Confidence Interval); unit: Probability of Event Free
Arm/Group | Overall Study
Number analyzed (Participants) | 166
Probability of Event Free
  12-Months Post-Index Procedure | 0.928 [0.878 to 0.958]
  24-Months Post-Index Procedure | 0.699 [0.619 to 0.765]

7. Secondary Outcome: Primary Target Lesion Patency (TLP) for Lesions > 160 mm at 12, 24, and 36 Months Post-Index Procedure
Description: Primary Target Lesion Patency (TLP) - Sustained and Expanded - for Target Lesion Lengths > 160 mm at 12-, 24- and 36-months post-index procedure corresponding to Peak Systolic Ratio (PSR) values of < 2.0, <2.5, and < 3.0.
Time Frame: 12, 24, and 36 months Post Index Procedure
Population: Eighteen (18) patients were enrolled with lesions >160mm, therefore N=18. However, 15 patients had available data for analysis at 12, 24 and 36 months, therefore n=15.
Measure: Number (90% Confidence Interval); unit: Probability of Event Free
Arm/Group | LifeStent
Number analyzed (Participants) | 18
Probability of Event Free
  At 12-months (PSR < 2.0): number analyzed (Participants) | 15
  At 12-months (PSR < 2.0) | 0.464 [0.234 to 0.667]
  At 24-months (PSR < 2.0): number analyzed (Participants) | 15
  At 24-months (PSR < 2.0) | 0.155 [0.037 to 0.349]
  At 36-months (PSR < 2.0): number analyzed (Participants) | 15
  At 36-months (PSR < 2.0) | 0.155 [0.037 to 0.349]
  At 12-months (PSR < 2.5): number analyzed (Participants) | 15
  At 12-months (PSR < 2.5) | 0.464 [0.234 to 0.667]
  At 24-months (PSR < 2.5): number analyzed (Participants) | 15
  At 24-months (PSR < 2.5) | 0.232 [0.076 to 0.438]
  At 36-months (PSR < 2.5): number analyzed (Participants) | 15
  At 36-months (PSR < 2.5) | 0.232 [0.076 to 0.438]
  At 12-months (PSR < 3.0): number analyzed (Participants) | 15
  At 12-months (PSR < 3.0) | 0.464 [0.234 to 0.667]
  At 24-months (PSR < 3.0: number analyzed (Participants) | 15
  At 24-months (PSR < 3.0 | 0.232 [0.076 to 0.438]
  At 36-months (PSR < 3.0): number analyzed (Participants) | 15
  At 36-months (PSR < 3.0) | 0.232 [0.076 to 0.438]

8. Secondary Outcome: Freedom From Target Lesion Revascularization (TLR) and/or Target Vessel Revascularization (TVR) at 12, 24, and 36-Months Post-Index Procedure for Target Lesion Lengths > 160 mm.
Description: Freedom from Target Lesion Revascularization (TTR) and/or Target Vessel Revascularization (TRV) for Target Lesion Lengths > 160 mm at 12-, 24- and 36-months post-index procedure.
Time Frame: 12-, 24-, and 36-months post-index procedure
Measure: Number (90% Confidence Interval); unit: Probability of Event Free
Arm/Group | LifeStent
Number analyzed (Participants) | 173
Probability of Event Free
  12-months post-index procedure | 0.696 [0.436 to 0.854]
  24-months post-index procedure | 0.696 [0.436 to 0.854]
  36-months post index procedure | 0.696 [0.436 to 0.854]

9. Secondary Outcome: Secondary Safety Endpoint: Freedom From Composite Adverse Events
Description: Secondary Safety (Freedom from Composite Adverse Events) is defined as freedom from death (excluding 30-days and 12-months post-index procedure), stroke, myocardial infarction (MI), emergent surgical revascularization, significant distal embolization in target limb, target limb major amputation, and thrombosis of target vessel at 30-days and 12-, 24-, and 36-months post-index procedure.
Time Frame: 30-days and 12-, 24-, and 36-months post-index procedure
Population: (n) varies in relation to the number of evaluable subjects at 30 days, 12, 24, and 36 months. Accordingly, the (n) for each period may be different from the overall (N) reported in the Participant Flow section
Measure: Number (90% Confidence Interval); unit: Probability of Event Free
Arm/Group | LifeStent
Number analyzed (Participants) | 173
Probability of Event Free
  30-days Post Index Procedure: number analyzed (Participants) | 167
  30-days Post Index Procedure | 0.994 [0.970 to 0.999]
  12-Months Post Index Procedure: number analyzed (Participants) | 148
  12-Months Post Index Procedure | 0.988 [0.961 to 0.996]
  24-Months Post-Index Procedure: number analyzed (Participants) | 119
  24-Months Post-Index Procedure | 0.945 [0.904 to 0.969]
  36-Months Post-Index Procedure: number analyzed (Participants) | 67
  36-Months Post-Index Procedure | 0.901 [0.847 to 0.936]

10. Secondary Outcome: Number of Stents Deployed With Acute Technical Success
Description: Acute technical success is defined as successful deployment of the stent to the intended location.
Time Frame: Intra-procedure
Measure: Count of Units; unit: Stents
Units Other Than Participants: Stents
Arm/Group | LifeStent
Number analyzed (Participants) | 173
Number analyzed (Stents) | 217
Stents | 201

11. Secondary Outcome: Number of Acute Lesion Success
Description: Acute lesion success is defined as attainment of ≤ 30% residual stenosis of the target lesion using any percutaneous method and/or non-investigational device (i.e., post-dilatation) based on angiographic data.
Time Frame: Intra-procedure
Population: N=175 (lesions) differs from the baseline characteristics module that mentions 187 treated lesions due to availability of angiographic image that show less than, or equal to 30% residual stenosis post-dilatation, as evaluated by the independent core-lab at time of analysis.
Measure: Count of Units; unit: Target lesions
Units Other Than Participants: Target lesions
Arm/Group | LifeStent
Number analyzed (Participants) | 173
Number analyzed (Target lesions) | 175
Target lesions | 152

12. Secondary Outcome: Number of Procedures With Acute Success
Description: Acute procedure success is defined as lesion success and no peri-procedural complications (death, stroke, MI, emergent surgical revascularization, significant distal embolization in target limb, and thrombosis of target vessel).
Time Frame: Intra-procedure
Population: One patient died at day 22, therefore, in this analysis N=172 instead of N=173.
Measure: Count of Units; unit: Procedures
Units Other Than Participants: Procedures
Arm/Group | LifeStent
Number analyzed (Participants) | 172
Number analyzed (Procedures) | 172
Procedures | 149

13. Secondary Outcome: Sustained Freedom From Target Lesion Reintervention (TLR) and/or Target Vessel Reintervention (TVR) at 24 and 36 Months Post-Index Procedure
Description: Sustained Freedom from Target Lesion Reintervention (TLR) and/or Target Vessel Reintervention (TVR) at 24- and 36-months post-index procedure.
Time Frame: 24- and 36-months post-index procedure
Measure: Number (90% Confidence Interval); unit: Probability of Freedom from TLR or TRV
Arm/Group | LifeStent
Number analyzed (Participants) | 173
Probability of Freedom from TLR or TRV
  24-Months Post-Index Procedure | 0.669 [0.600 to 0.729]
  36-Months Post-Index Procedure (PSR < 2.5) | 0.631 [0.560 to 0.695]

14. Secondary Outcome: Number of Participants With Sustained Hemodynamic Success at 30-days, 12-, 24-, and 36-Months Post Index Procedure
Description: Sustained hemodynamic success is defined as sustained improvement of Ankle-Brachial Index (ABI) from baseline value of ≥ 0.15 at 30-days and 12-, 24-, and 36-months post-index procedure without the need for repeated Target Lesion Revascularization (TLR) in surviving subjects.
Time Frame: 30 days, 12-, 24-, and 36-months post-index procedure
Population: The number of participants for each time period represents the evaluable subjects for this specific outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 99
Participants
  30-Days Post Index Procedure | 64
  12-Months Post-Index Procedure: number analyzed (Participants) | 85
  12-Months Post-Index Procedure | 32
  24-Months Post-Index Procedure: number analyzed (Participants) | 69
  24-Months Post-Index Procedure | 17
  36-Months Post-Index Procedure: number analyzed (Participants) | 57
  36-Months Post-Index Procedure | 13

15. Secondary Outcome: Number of Participants With Sustained Clinical Success at 30-Days, 12, 24, and 36- Months Post-Index Procedure
Description: Sustained clinical success is defined as sustained cumulative improvement from baseline value of ≥ 1 category according to Rutherford et al.12 at 30-days and 12-, 24-, and 36-months post-index procedure without the need for repeated TLR in surviving subjects.
Time Frame: 30-days and 12-, 24-, and 36-months post-index procedure
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 157
Participants
  30-days Post Index Procedure | 142
  12-Months Post Index Procedure: number analyzed (Participants) | 132
  12-Months Post Index Procedure | 91
  24-Months Post-Index Procedure: number analyzed (Participants) | 103
  24-Months Post-Index Procedure | 56
  36-Months Post-Index Procedure: number analyzed (Participants) | 78
  36-Months Post-Index Procedure | 33

16. Secondary Outcome: Sustained Target Lesion Patency (TLP) at 24 and 36 Months Post-Index Procedure
Description: Sustained Target Lesion Patency (TLP) was measured at 24- and 36-months post-index procedure corresponding to PSR < 2.5.
Time Frame: 24- and 36-months post-index procedure
Population: The results presented in this analysis include active patients that had available ultrasound images appropriate for analysis by the independent core-lab at follow-up time (24 and 36 months). Therefore n=161 instead of N=173.
Measure: Number (90% Confidence Interval); unit: Probability of sustained lesion patency
Arm/Group | Overall Study
Number analyzed (Participants) | 161
Probability of sustained lesion patency
  24-Months Post-Index Procedure (PSR < 2.5) | 0.510 [0.436 to 0.578]
  36-Months Post-Index Procedure (PSR < 2.5) | 0.457 [0.382 to 0.529]

17. Secondary Outcome: Expanded Target Lesion Patency (TLP) for Peak Systolic Velocity Ratio (PSR) < 3.0 at 12, 24, and 36 Months Post-Index Procedure
Description: Expanded TLP was measured at 12-, 24- and 36-months post-index procedure corresponding to Peak Systolic Velocity Ratio (PSR) < 3.0.
Time Frame: 12, 24, and 36 months Post-Index Procedure
Population: The results presented in this analysis include active patients that had available ultrasound images appropriate for analysis by the independent core-lab at follow-up time (12, 24 and 36 months). Therefore n=161 instead of N=173.
Measure: Number (90% Confidence Interval); unit: Probability of Lesion Patency
Units Other Than Participants: Lesion
Arm/Group | LifeStent
Number analyzed (Participants) | 161
Number analyzed (Lesion) | 161
Probability of Lesion Patency
  At 12-months (PSR < 3.0) | 0.761 [0.696 to 0.814]
  At 24-months (PSR < 3.0) | 0.523 [0.450 to 0.591]
  At 36-months (PSR < 3.0) | 0.470 [0.394 to 0.542]

18. Secondary Outcome: Cumulative (Primary Assisted and Secondary) Target Lesion Patency (TLP) at 12, 24, and 36 Months Post-Index Procedure
Description: Cumulative (primary-assisted and secondary) Target Lesion Patency (TLP) was measured at 12-, 24-, and 36-months post-index procedure corresponding to Peak Systolic Velocity Ratio (PSR) < 2.5, and PSR < 3.0.
Time Frame: 12, 24, and 36 Months Post-Index Procedure
Population: The results presented in this analysis include active patients that had available ultrasound images appropriate for analysis by the independent core-lab at follow-up time (12, 24 and 36 months). Therefore n=160 instead of N=173.
Measure: Number (90% Confidence Interval); unit: Probability of Target Lesion Patency
Units Other Than Participants: Lesions
Arm/Group | LifeStent
Number analyzed (Participants) | 160
Number analyzed (Lesions) | 160
Probability of Target Lesion Patency
  At 12-months (PSR < 2.5) | 0.920 [0.873 to 0.951]
  At 24-months (PSR < 2.5) | 0.745 [0.675 to 0.802]
  At 36-months (PSR < 2.5) | 0.717 [0.644 to 0.777]
  At 12-months (PSR < 3.0) | 0.928 [0.882 to 0.956]
  At 24-months (PSR < 3.0) | 0.784 [0.717 to 0.837]
  At 36-months (PSR < 3.0) | 0.745 [0.673 to 0.803]

19. Secondary Outcome: Change From Baseline in Walking Impairment Questionnaire (WIQ) Results at 30-Days and 12, 24 and 36-Months Post-Index Procedure
Description: The Walking Impairment Questionnaire (WIQ) evaluation scale values range from 0 to 100, with 0 meaning inability to complete the specific task and 100 representing no difficulty in completing the task. A higher score (mean) represents an improvement in walking abilities compared to baseline measure. The results below represent, for each item measured (pain, walking distance, walking speed, and stair climbing), the mean difference between the score observed at Baseline and those observed at 30-days, 12-, 24-, and 36-months post-index procedure.
Time Frame: 30-days, and 12-, 24-, and 36-months post-index procedure
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Overall Study
Number analyzed (Participants) | 159
Score on a Scale
  Pain at 30-days Post-Index Procedure: number analyzed (Participants) | 145
  Pain at 30-days Post-Index Procedure | 43.4 (34.61)
  Pain at 12-Months Post-Index Procedure: number analyzed (Participants) | 129
  Pain at 12-Months Post-Index Procedure | 30.8 (39.59)
  Pain at 24-Months Post-Index Procedure: number analyzed (Participants) | 102
  Pain at 24-Months Post-Index Procedure | 33.8 (42.46)
  Pain at 36-Months Post-Index Procedure: number analyzed (Participants) | 74
  Pain at 36-Months Post-Index Procedure | 30.7 (40.24)
  Walking Distance at 30-days Post-Index Procedure: number analyzed (Participants) | 147
  Walking Distance at 30-days Post-Index Procedure | 26.46 (33.55)
  Walking Distance at 12-Months Post-Index Procedure: number analyzed (Participants) | 130
  Walking Distance at 12-Months Post-Index Procedure | 19.89 (35.83)
  Walking Distance at 24-Months Post-Index Procedure: number analyzed (Participants) | 103
  Walking Distance at 24-Months Post-Index Procedure | 22.97 (30.83)
  Walking Distance at 36-Months Post-Index Procedure: number analyzed (Participants) | 76
  Walking Distance at 36-Months Post-Index Procedure | 26.39 (35.99)
  Walking Speed at 30-days Post-Index Procedure: number analyzed (Participants) | 146
  Walking Speed at 30-days Post-Index Procedure | 18.09 (24.51)
  Walking Speed at 12-Months Post-Index Procedure: number analyzed (Participants) | 129
  Walking Speed at 12-Months Post-Index Procedure | 13.39 (27.23)
  Walking Speed at 24-Months Post-Index Procedure: number analyzed (Participants) | 103
  Walking Speed at 24-Months Post-Index Procedure | 14.64 (23.37)
  Walking Speed at 36-Months Post-Index Procedure: number analyzed (Participants) | 76
  Walking Speed at 36-Months Post-Index Procedure | 13.19 (27.33)
  Stair Climbing at 30-days Post-Index Procedure: number analyzed (Participants) | 141
  Stair Climbing at 30-days Post-Index Procedure | 22.19 (34.37)
  Stair Climbing at 12-Months Post-Index Procedure: number analyzed (Participants) | 126
  Stair Climbing at 12-Months Post-Index Procedure | 16.96 (34.80)
  Stair Climbing at 24-Months Post-Index Procedure: number analyzed (Participants) | 99
  Stair Climbing at 24-Months Post-Index Procedure | 16.96 (34.81)
  Stair Climbing at 36-Months Post-Index Procedure: number analyzed (Participants) | 73
  Stair Climbing at 36-Months Post-Index Procedure | 10.05 (38.47)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment until final patient follow up visit (36-months follow up or end of study visit).
Arm/Group | LifeStent
All-Cause Mortality (participants affected / at risk) | 22/173
Serious Adverse Events (participants affected / at risk) | 111/173
Other Adverse Events (participants affected / at risk) | 150/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LifeStent (N=173)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 6 (6)
Angina pectoris (Cardiac disorders) | 7 (7)
Angina unstable (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 4 (4)
Cardiac failure acute (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 11 (11)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 9 (9)
Coronary artery stenosis (Cardiac disorders) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (8)
Haematemesis (Gastrointestinal disorders) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Chest pain (General disorders) | 3 (3)
Device breakage (General disorders) | 2 (2)
Device dislocation (General disorders) | 1 (1)
Device occlusion (General disorders) | 2 (2)
Granuloma (General disorders) | 1 (1)
Ischaemic ulcer (General disorders) | 2 (2)
Medical device complication (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Ulcer (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 7 (7)
Clostridial infection (Infections and infestations) | 2 (2)
Diabetic foot infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Furuncle (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 2 (2)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Postoperative wound infection (Infections and infestations) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Septic shock (Infections and infestations) | 1 (1)
Serratia infection (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (7)
Viral pericarditis (Infections and infestations) | 1 (1)
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 4 (4)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1)
Positron emission tomogram abnormal (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 4 (4)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 5 (5)
Convulsion (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Neuromyopathy (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 4 (4)
Transient ischaemic attack (Nervous system disorders) | 4 (4)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 3 (3)
Renal failure chronic (Renal and urinary disorders) | 3 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3)
Angioplasty (Surgical and medical procedures) | 1 (1)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 2 (2)
Coronary artery bypass (Surgical and medical procedures) | 1 (1)
Gastric tube reconstruction (Surgical and medical procedures) | 1 (1)
Peripheral artery angioplasty (Surgical and medical procedures) | 1 (1)
Peripheral revascularisation (Surgical and medical procedures) | 1 (1)
Polypectomy (Surgical and medical procedures) | 1 (1)
Vascular operation (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Arterial stenosis limb (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Carotid artery stenosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 6 (6)
Femoral arterial stenosis (Vascular disorders) | 5 (5)
Femoral artery occlusion (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 16 (16)
Ischaemia (Vascular disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 9 (9)
Peripheral ischaemia (Vascular disorders) | 4 (4)
Peripheral vascular disorder (Vascular disorders) | 16 (16)
Venous insufficiency (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LifeStent (N=173)
Anemia (Blood and lymphatic system disorders) | 20 (20)
Angina pectoris (Cardiac disorders) | 11 (11)
Cardiac failure congestive (Cardiac disorders) | 14 (14)
Coronary artery disease (Cardiac disorders) | 10 (10)
Device breakage (General disorders) | 12 (12)
Oedema peripheral (General disorders) | 12 (12)
Cellulitis (Infections and infestations) | 14 (14)
Pneumonia (Infections and infestations) | 11 (11)
Urinary tract infection (Infections and infestations) | 17 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 (23)
Neuropathy peripheral (Nervous system disorders) | 9 (9)
Renal failure acute (Renal and urinary disorders) | 17 (17)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Femoral artery stenosis (Vascular disorders) | 10 (10)
Haematoma (Vascular disorders) | 14 (14)
Intermittent claudication (Vascular disorders) | 25 (25)
Peripheral arterial occlusive disease (Vascular disorders) | 15 (15)
Peripheral vascular disorder (Vascular disorders) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to PI publication of site results, sponsor requires publication of multi-centers results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT00908947/Prot_SAP_000.pdf